CLINICAL TRIAL: NCT03315975
Title: Influenza Vaccine Responses in the Setting of Melanoma Treatment
Brief Title: Flu Vaccine Responses in the Setting of Melanoma Treatment
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 826207
Record Dates: First submitted 2017-10-16; First posted 2017-10-20 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Viral Vaccines
Keywords: Influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Influenza vaccination cohort (Experimental): Subjects will receive one dose of seasonal quadrivalent inactivated influenza vaccine intramuscularly for standard of care for prevention of influenza infection.
  Interventions: Biological: Inactivated influenza vaccine

INTERVENTIONS:
Biological: Inactivated influenza vaccine — One dose of quadrivalent inactivated influenza vaccine

SUMMARY:
Influenza vaccination is indicated for all adults, but the immunogenicity of vaccination has not been assessed in all situations. We are conducting a prospective unblinded study of influenza vaccine recipients.

DETAILED DESCRIPTION:
Influenza vaccination is indicated for all adults, but the immunogenicity of vaccination has not been assessed in all situations. In particular, immune responses following influenza vaccination have not been studied in the setting of advanced melanoma and in the context of various anti-tumor treatments. In this study, we will look at the immune response of subjects receiving vaccination.

ELIGIBILITY:
Inclusion Criteria:

* adults capable of providing consent
* have a diagnosis of locally advanced or metastatic melanoma

Exclusion Criteria:

* are allergic to influenza vaccination
* have received influenza vaccination within the past 6 months
* require prednisone, methotrexate, or other immunosuppressing medications
* have HIV infection
* have a history of solid organ or bone marrow transplant
* require combination immunotherapy
* are on other studies requiring blood draws that might exceed 450 mL total during the period of the influenza vaccine study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-10-20 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Neutralizing antibody response | 21-42 days
  The neutralizing antibody titer will be assessed by measurement of the hemagglutinin-inhibition titer before and after influenza vaccination in order to determine the seroconversion rate. The late blood draw may occur between days 21-42 following vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: E. John Wherry, PhD, Principal Investigator — University of Pennsyvlania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No